CLINICAL TRIAL: NCT01914159
Title: Ranibizumab In Pigment Epithelium Tears Secondary To Age-Related Macular Degeneration Study
Acronym: RIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Frank G. Holz, Director, Department of Ophthalmology, University of Bonn, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-037.0156
Record Dates: First submitted 2013-07-28; First posted 2013-08-01 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab (Lucentis, Novartis Pharma GmbH, Germany)

INTERVENTIONS:
Drug: Ranibizumab (Lucentis, Novartis Pharma GmbH, Germany) — Monthly intravitreal injections

SUMMARY:
The Ranibizumab in Pigment Epithelium Tears Secondary To Age-Related Macular Degeneration (RIP) Study is a prospective, multicenter, uncontrolled, interventional phase 2 clinical trial that investigates the effect of fixed monthly intravitreal injections of ranibizumab (Lucentis, Novartis Pharma, Germany) on visual acuity and retinal morphology over a study period of 12 months in 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a pigment epithelial tear secondary to age-related macular degeneration
* Written informed consent

Exclusion Criteria:

* Time of diagnosis more than 6 months before study recruitment
* Ocular surgery of the study eye within 1 month before study recruitment
* Extensive subretinal fibrosis or retinal atrophy of the study eye
* Significant opacification of optical media of the study eye
* Uncontrolled glaucoma of the study eye
* Active ocular inflammation of the study eye
* Best-corrected visual acuity of the contralateral eye below 20/200
* Concurrent ocular or systemic therapy with other vascular endothelial growth factor (VEGF)-inhibitory drugs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University of Bonn, Department of Ophthalmology, Bonn
  - University of München (LMU), Department of Ophthalmology, München
  - Universityof Münster, Department of Ophthalmology, Münster

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab
Started | 24
Completed | 21
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 24
Best-corrected visual acuity [Mean (Standard Deviation); unit: ETDRS letters] | 50.3 (18.7)
Central retinal thickness [Mean (Standard Deviation); unit: µm] | 571 (185)
Vision-related quality of life [Mean (Standard Deviation); unit: NEI VFQ-25 score] — National Eye Institute Visual Function Questionaire 25-item version (NEI VFQ-25)
  0 to 100 scale, where 100 represents the best possible score and 0 represents the worst
  Reference: Mangione CM et al. Arch Ophthalmol 2001 Jul;119(7):1050-8.
  NEI VFQ-25 score | 79.0 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Best-corrected Visual Acuity
Description: Early Treatment of Diabetic Retinopathy Study (ETDRS) protocol
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 24
ETDRS letters | 52.9 (19.7)

2. Secondary Outcome: Retinal Morphology
Description: Spectral-domain optical coherence tomography (SD-OCT) central retinal thickness
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab
Number analyzed (Participants) | 24
µm | 436 (171)

3. Secondary Outcome: Vision-related Quality of Life
Description: National Eye Institute Visual Function Questionaire 25-item version (NEI VFQ-25)
  0 to 100 scale, where 100 represents the best possible score and 0 represents the worst
  Reference: Mangione CM et al. Arch Ophthalmol 2001 Jul;119(7):1050-8.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: NEI VFQ-25 score
Arm/Group | Ranibizumab
Number analyzed (Participants) | 24
NEI VFQ-25 score | 74.3 (13.9)

ADVERSE EVENTS:
Arm/Group | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab (N=24)
Increase of subretinal hemorrhage (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes